CLINICAL TRIAL: NCT01383954
Title: The Efficacy of Diclofenac Gel for Breakthrough Pain and the Neuropathic Components of Pain in Knee Osteoarthritis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Endo Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Ajay D. Wasan,M.D.,M.Sc., Investigator, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2009p000667
Record Dates: First submitted 2011-06-22; First posted 2011-06-28 (Estimated); Results first posted 2017-07-06 (Actual); Last update posted 2017-08-15 (Actual); Status verified 2017-07

CONDITIONS: Knee Osteoarthritis
Keywords: Knee osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Diclofenac

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Diclofenac gel (Other): Diclofenac gel 4 grams (g) applied topically 4 times daily (QID) to the affected knee(s) for up to 4 weeks. Participants took a maximum dosage of 32 g/day.
  Interventions: Drug: Diclofenac Gel

INTERVENTIONS:
Drug: Diclofenac Gel — Diclofenac gel 4 grams (g) applied topically 4 times daily (QID) to the affected knee(s) for up to 4 weeks. Participants took a maximum dosage of 32 g/day.
  Other Names: Voltaren

SUMMARY:
The purpose of this proposed study is to conduct a trial with knee osteoarthritis (OA) patients using the diclofenac gel.

DETAILED DESCRIPTION:
The purpose of this proposed study is to conduct a trial with knee OA patients using the diclofenac gel. The effectiveness of diclofenac gel in managing breakthrough pain or the neuropathic components of pain (e.g., the burning, soft tissue joint sensitivity, or allodynic components) in knee OA is unknown. It is likely that patients will use the gel in a as needed (prn) fashion, on top of other analgesics prescribed for their pain. The neuropathic components of a generally nociceptive or inflammatory condition, such as knee OA, are underappreciated, and typically not tracked in OA analgesic studies. Yet, evidence across a variety of chronic painful conditions suggests that these components are quite disabling. The results of this study would show whether diclofenac gel as a prn medication is beneficial to patients suffering from knee OA pain.

ELIGIBILITY:
Inclusion Criteria:

* Ages 20-75
* Unilateral or bilateral knee osteoarthritis (OA), confirmed radiographically.
* Patients taking oral non-steroidal anti-inflammatory drugs (NSAIDs) in the amount and schedule prior to the breakthrough period will be permitted.

Exclusion Criteria:

* Patients with clinical history of anterior cruciate ligament (ACL) involvement.
* Patients on tricyclic antidepressants or anticonvulsants (neuropathic medications)
* History of ulcers or gastrointestinal (GI) bleeding
* Coagulation disorders
* Hypersensitivity to Aspirin or NSAIDS
* Congestive Heart Failure and Edema
* Advanced renal disease
* Aspirin triad
* Pregnant women

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2011-06 (Actual); Primary Completion 2012-08 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ajay D Wasan, M.D, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Chestnut Hill, Massachusetts, United States

REFERENCES:
- [Derived] Edwards RR, Dolman AJ, Martel MO, Finan PH, Lazaridou A, Cornelius M, Wasan AD. Variability in conditioned pain modulation predicts response to NSAID treatment in patients with knee osteoarthritis. BMC Musculoskelet Disord. 2016 Jul 13;17:284. doi: 10.1186/s12891-016-1124-6. PMID 27412526

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Diclofenac Gel
Started | 52
Safety Population: Received Treatment | 48
Completed (Completed = completed at least 2 weeks of being on study medication) | 38
Not Completed | 14
Not completed — Lack of Efficacy | 2
Not completed — Electronic Diary Too Cumbersome to Use | 2
Not completed — Adverse Event | 1
Not completed — Reason Not Specified | 9

BASELINE CHARACTERISTICS:
Population: Modified Intent-to-Treat Population, all participants who completed at least 50% of the study (at least 2 weeks of drug treatment).
Arm/Group | Diclofenac Gel
Number analyzed (Participants) | 38
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.8 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 15

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Pain Score During Week 1
Description: Participants assessed their knee pain using a visual analog scale (VAS) where 0=no pain and 100=worst possible pain. Pain scores were recorded in an electronic diary prior to and 4 hours after the first daily application of diclofenac gel for breakthrough pain. The daily percent change in pain scores over the 7 days prior to Week 1 were averaged. Percent change from Baseline (average pain score 7 days prior to first treatment) was calculated as (value at baseline - value at post-baseline visit) / (value at baseline) x 100. A positive change from Baseline indicates improvement.
Time Frame: Baseline and Week 1
Population: Modified Intent-to-Treat Population, all participants who completed at least 50% of the study (at least 2 weeks of drug treatment), who had pain data available for analysis at the given timepoints.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Diclofenac Gel
Number analyzed (Participants) | 38
percent change | 33.3 (23.7)

2. Primary Outcome: Percent Change From Baseline in Pain Score During Week 2
Description: Participants assessed their knee pain using a visual analog scale (VAS) where 0=no pain and 100=worst possible pain. Pain scores were recorded in an electronic diary prior to and 4 hours after the first daily application of diclofenac gel for breakthrough pain. The daily percent change in pain scores over the 7 days prior to Week 2 were averaged. Percent change from baseline (average pain score 7 days prior to first treatment) was calculated as (value at baseline - value at post-baseline visit)/ (value at baseline) x 100. A positive change from baseline indicates improvement.
Time Frame: Baseline and Week 2
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Diclofenac Gel
Number analyzed (Participants) | 37
percent change | 33.3 (23.7)

ADVERSE EVENTS:
Arm/Group | Diclofenac Gel
Serious Adverse Events (participants affected / at risk) | 0/48
Other Adverse Events (participants affected / at risk) | 1/48
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Diclofenac Gel (N=48)
Rash (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes